CLINICAL TRIAL: NCT02031939
Title: Randomized Controlled Study on Optimize Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Hai Lu, Pofessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013013; SYSU5010Fund (Other Grant/Funding Number: Sun Yat-Sen University 5010 Fund)
Record Dates: First submitted 2013-12-30; First posted 2014-01-09 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Advanced Rectal Cancer
Keywords: Rectal cancer; neoadjuvant chemoradiotherapy; optimization
MeSH Terms: conditions — Rectal Neoplasms | interventions — Induction Chemotherapy; Chemoradiotherapy; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard chemoradiotherapy (Active Comparator): Standard chemoradiotherapy (Capecitabine 825mg/m2 combined with radiotherapy )
  Interventions: Radiation: standard chemoradiotherapy
- induction and gap chemotherapy (Experimental): induction chemotherapy (Capecitabine 2000mg/m2 +oxaliplatine 130mg/m2) + 2 cycles of chemoradiotherapy (Capecitabine 2000mg/m2 +oxaliplatine 100mg/m2 combined with radiotherapy) + gap chemotherapy (Capecitabine 2000mg/m2 + oxaliplatine 130mg/m2)
  Interventions: Drug: Induction chemotherapy, Chemoradiotherapy and gap chemotherapy (Capecitabine combine with oxaliplatin)

INTERVENTIONS:
Drug: Induction chemotherapy, Chemoradiotherapy and gap chemotherapy (Capecitabine combine with oxaliplatin) — All rectal cancer patients in this group will receive induction, gap chemotherapy (capecitabine combined with oxaliplatin) alone with chemoradiotherapy (capecitabine combine with oxaliplatin) before surgery.
  Arms: induction and gap chemotherapy
Radiation: standard chemoradiotherapy — All rectal patients in this group will receive standard radiotherapy and surgical resection.
  Arms: Standard chemoradiotherapy

SUMMARY:
Although neoadjuvant chemoradiotherapy has significantly reduced the risk of local recurrence in locally advanced rectal cancer, systemic failure remains a predominant issue probably due to the insufficient control of systemic micro-metastasis in the neoadjuvant treatment. Induction chemotherapy is one of the most studied strategies. However, the efficacy of induction chemotherapy prior to neoadjuvant chemotherapy remains controversial. In our previous study, induction chemotherapy, gap chemotherapy combined with neoadjuvant chemoradiotherapy can improve response rate of rectal cancer patients, but the results have not been confirmed in clinical trial. Whether this new kind of treatment can optimize neoadjuvant therapy for locally advanced rectal cancer or not is still a big problem in clinical practice. This study will focus on how to optimize neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed rectal cancer
* Clinical stage T3-4 or T any N1
* No metastasis
* Distance of tumor is no more than 10cm from anal verge
* No previous radiotherapy
* Age ranged from 18 to 70
* Eastern Cooperative Oncology Group score system 0-1

Exclusion Criteria:

* Clinical stage T1-2 N0
* Distance metastasis
* Multiple primary tumor
* Cachexy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years

SECONDARY OUTCOMES:
disease free survival | 3 years
Disease free survival | 5 years
Respond rate | One week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Hai Lu, Prof., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China